CLINICAL TRIAL: NCT04984525
Title: A Phase 1, Dose-escalation, Placebo- and Active-Controlled Crossover Study to Assess the Safety, Tolerability, and Pharmacodynamics of SYNB1934 and the Effect of Concomitant Proton Pump Inhibitor Administration in Healthy Volunteers
Brief Title: Safety and Tolerability of SYNB1934 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synlogic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SYNB1934-CP-001
Record Dates: First submitted 2021-07-21; First posted 2021-07-30 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Part 1:
  Triple (Participant, Care Provider, Investigator) Double-blind (Sponsor-open)
  Part 2:
  Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1 Cohort 1 MAD HV: SYNB1934 (3 x 10^11 live cells) (Experimental): HV subjects receive SYNB1934 (3 x 10^11 live cells) At least 3 times per day (TID) on Treatment Day 1 and once at breakfast on Treatment Day 2
  Interventions: Drug: SYNB1934
- Part 1 Cohort 2 Crossover HV: SYNB1934 (6 x 10^11 live cells) (Experimental): HV subjects receive SYNB1934 (6 x 10^11 live cells) At least 3 times per day (TID) on Treatment Day 1 and once at breakfast on Treatment Day 2 Following a ≥ 7-day washout period HV subjects receive SYNB1618 (6 x 10^11 live cells), at least 3 times per day (TID) on Treatment Day 1 and once at breakfast on Treatment Day 2
  Interventions: Drug: SYNB1934; Drug: SYNB1618
- Part 1 Cohort 3 MAD HV: SYNB1934 (1 x 10^12 live cells) (Experimental): HV subjects receive SYNB1934 (1 x 10^12 live cells) At least 3 times per day (TID) on Treatment Day 1 and once at breakfast on Treatment Day 2
  Interventions: Drug: SYNB1934
- Part 1 Cohort 4 MAD HV: SYNB1934 (optional) (Experimental): HV subjects receive SYNB1934 (at a dose to be determined based on the data from the first 3 cohorts) At least 3 times per day (TID) on Treatment Day 1 and once at breakfast on Treatment Day 2
  Interventions: Drug: SYNB1934
- Part 1 Cohort 5 MAD HV: SYNB1934 (optional) (Experimental): HV subjects receive SYNB1934 (at a dose to be determined based on the data from the first 3 cohorts) At least 3 times per day (TID) on Treatment Day 1 and once at breakfast on Treatment Day 2
  Interventions: Drug: SYNB1934
- Part 2 Crossover with PPI vs No PII (Experimental): HV subjects receive SYNB1934 (at or below the MTD from Part 1) with PPI At least 3 times per day (TID) on Treatment Day 1 and once at breakfast on Treatment Day 2 Following a ≥ 14-day washout period HV subjects receive SYNB1934 (at or below the MTD from Part 1) without PPI At least 3 times per day (TID) on Treatment Day 1 and once at breakfast on Treatment Day 2
  Interventions: Drug: SYNB1934

INTERVENTIONS:
Drug: SYNB1934 — SYNB1934 is formulated as a nonsterile solution intended for oral administration
Drug: SYNB1618 — SYNB1618 is formulated as a nonsterile solution intended for oral administration
  Arms: Part 1 Cohort 2 Crossover HV: SYNB1934 (6 x 10^11 live cells)

SUMMARY:
This Phase 1, first-in-human, multiple dose-escalation, randomized, double-blinded, placebo-controlled study is evaluating SYNB1934 in healthy volunteers (HV). Eligible subjects receive investigational product (IP) and undergo safety monitoring, evaluations, and subsequent follow-up after IP administration.

DETAILED DESCRIPTION:
This study is evaluating the safety, tolerability, kinetics, and pharmacodynamics of SYNB1934 within the following 2 study parts:

Part 1 is an inpatient, placebo-controlled, multiple ascending dose (MAD) study in HV male and female subjects in up to 5 dose cohorts (6 treated: 2 placebo) for 5 days of dosing to identify the maximum tolerated dose (MTD). During the second cohort an additional 6 treated subjects will be enrolled; all treated subjects in Cohort 2 will complete a second treatment period with SYNB1618 in a cross-over design.

Part 2 is an open-label, randomized sequence, crossover study of SYNB1934 that will be initiated after determination and selection of a well-tolerated dose in Part 1. Subjects will receive treatment with SYNB1934 with a proton pump inhibitor (PPI), will complete a treatment washout period, and receive SYNB1934 treatment without a PPI. Initially 16 HV male and female subjects will be enrolled with the option of expanding Part 2 up to 60 HV subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 to ≤ 64 years.
2. Able and willing to voluntarily complete the informed consent process.
3. Available for and agree to all study procedures, including feces, urine, and blood collection and adherence to diet control, inpatient monitoring, follow-up visits, and compliance with all study procedures.
4. Male subjects who are sexually abstinent or surgically sterilized (vasectomy), or those who are sexually active with a female partner(s) and agree to use an acceptable method of contraception (such as a condom with spermicide) combined with an acceptable method of contraception for their non-pregnant female partner(s) (as defined in Inclusion Criterion # 5) after informed consent, throughout the study, and for a minimum of 3 months after the last dose of IMP, and who do not intend to donate sperm in the period from Screening until 3 months following administration of the IMP.
5. Female subjects who meet 1 of the following:

   1. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (human chorionic gonadotropin) at Screening and a negative urine pregnancy test at baseline prior to the start of IMP and must agree to use acceptable method(s) of contraception, combined with an acceptable method of contraception for their male partner(s) (as defined in Inclusion Criterion # 4) after informed consent, throughout the study and for a minimum of 3 months after the last dose of IMP. Acceptable methods of contraception include hormonal contraception, hormonal or non-hormonal intrauterine device, bilateral tubal occlusion, complete abstinence, vasectomized partner with documented azoospermia 3 months after procedure, diaphragm with spermicide, cervical cap with spermicide, vaginal sponge with spermicide, or male or female condom with or without spermicide.
   2. Premenopausal women with at least 1 of the following:

   i. Documented hysterectomy ii. Documented bilateral salpingectomy iii. Documented bilateral oophorectomy iv. Documented tubal ligation/occlusion v. Sexual abstinence is preferred or usual lifestyle of the subject

   c. Postmenopausal women (12 months or more amenorrhea verified by follicle-stimulating hormone assessment and over 45 years of age in the absence of other biological or physiological causes).

Exclusion Criteria:

1. Acute or chronic medical (including COVID-19 infection), surgical, psychiatric, or social condition or laboratory abnormality that may increase subject risk associated with study participation, compromise adherence to study procedures and requirements, or may confound interpretation of study safety or PD results and, in the judgment of the investigator, would make the subject inappropriate for enrollment.
2. Body mass index < 18.5 or ≥ 35 kg/m2.
3. History of or current immunodeficiency disorder including human immunodeficiency virus (HIV) antibody positivity.
4. Hepatitis B surface antigen positivity (subjects with hepatitis B surface antibody positivity and hepatitis B core antibody positivity are not excluded, provided that the hepatitis B surface antigen is negative).
5. Hepatitis C antibody positivity, unless a hepatitis C virus ribonucleic acid test is performed, and the result is negative.
6. History of febrile illness, confirmed bacteremia, or other active infection deemed clinically significant by the investigator within 30 days prior to the anticipated first dose of IMP.
7. History of (within the past month) passage of 3 or more loose stools per day, where "loose stool" is defined as a Type 6 or Type 7 on the Bristol Stool Chart.
8. Inflammatory or irritable bowel disorder of any grade experienced within the previous 60 days.
9. Active or past history of gastrointestinal bleeding within 60 days prior to the Screening Visit as confirmed by hospitalization-related event(s) or medical history of hematemesis or hematochezia.
10. Intolerance of or allergic reaction to EcN, esomeprazole, or any of the ingredients in SYNB1934 or placebo formulations. (For subjects who may be randomized to receive SYNB1618, intolerance of or allergic reaction to any of the ingredients in the SYNB1618 formulation.)
11. Any condition (e.g., celiac disease, gastrectomy, bypass surgery, ileostomy), prescription medication, or over-the-counter product that may possibly affect absorption of medications or nutrients.
12. Currently taking or plans to take any type of systemic (e.g., oral or intravenous) antibiotic within 30 days prior to Day -1 through the final day of inpatient monitoring. Exception: topical antibiotics are allowed.
13. Major surgery (an operation upon an organ within the cranium, chest, abdomen, or pelvic cavity) or inpatient hospital stay within the past 3 months prior to Screening.
14. Planned surgery, hospitalizations, dental work, or interventional studies between Screening and last anticipated visit.
15. Taking or planning to take probiotic supplements (enriched foods excluded) within 30 days prior to Day -1 through the Safety Follow-up Period.
16. Dependence on alcohol or drugs of abuse.
17. Administration or ingestion of an investigational drug within 30 days or 5 half-lives, whichever is longer, prior to the Screening Visit, or current enrollment in an investigational study.
18. Receipt of a COVID-19 vaccine 7 days prior to the anticipated first dose of IMP or 7 days after the last dose of IMP is permitted; otherwise, COVID-19 vaccines are not permitted during study participation.
19. Administration or ingestion of a PPI within 30 days prior to Day -2.
20. Screening laboratory parameters (e.g., chemistry panel, hematology, coagulation) and ECG outside of the normal limits based on standard ranges, or as judged to be clinically significant by the investigator. A single repeat evaluation is acceptable.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Number of Subjects With Treatment-Emergent Adverse Events | 70 days
  Toxicity is graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Adverse events (AEs) are reported based on clinical laboratory tests, vital signs, physical examinations, electrocardiograms, and any other medically indicated assessments from the time informed consent is signed through the end of the safety follow-up period.
  AEs are considered to be treatment emergent (TEAE) if they occur or worsen in severity after the first dose of study treatment. TEAEs are considered treatment-related if relationship to study drug is possibly related, probably related, or definitely related.

CONTACTS AND LOCATIONS:
Locations (1):
- High Point Clinical Trials Center, High Point, North Carolina, United States